CLINICAL TRIAL: NCT00692614
Title: A Phase IIb, Randomized, Masked, Sham-Controlled, Clinical Trial to Study the Efficacy and Safety of the Helical Triamcinolone Acetonide Implant (MK0140) in Diabetic Patients With Clinically Significant Macular Edema
Brief Title: A Study of MK0140 in Diabetic Patients With Macular Edema (0140-001)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0140-001; MK0140-001; 2008_521
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- 1 (Experimental): 100 mcg triamcinolone acetonide
  Interventions: Drug: triamcinolone acetonide
- 2 (Experimental): 500 mcg triamcinolone acetonide
  Interventions: Drug: triamcinolone acetonide
- 3 (Experimental): 925 mcg triamcinolone acetonide
  Interventions: Drug: triamcinolone acetonide
- 4 (No Intervention): sham control - not implanted, no medication

INTERVENTIONS:
Drug: triamcinolone acetonide — 100 mcg; 500 mcg; 925 mcg triamcinolone acetonide on helical coil implant to elute over 12 months.
  Other Names: MK0140
  Arms: 1; 2; 3

SUMMARY:
This study will evaluate the treatment effect of three doses of the I-vation TA implant (MK0140) in diabetic patients with clinically significant macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Patient has clinically significant macular edema as a result of their diabetes (Type I or Type 2)
* Patient has in the study eye, 20/40 - 20/160 vision
* Patient has Type 1 or Type 2 diabetes
* Patient agrees to remain abstinent or use (or have their partner use) 2 acceptable methods of birth control

Exclusion Criteria:

* Patient has had any active ocular infection in either eye
* Patient has intraocular pressure > 22 mmHg or a diagnosis of glaucoma
* Patient has cystoid macular edema in the study eye
* Patient has a history of elevated IOP in response to ocular steroid therapy in either eye
* Patient has had intraocular surgery in the study eye within 6 months prior to Visit 1
* Patient has an HbAIc value > 10% at Visit 1
* Patient has within the last 4 months initiated intensive insulin treatment or plan to do so in the next 4 months
* Patient has a history of cancer within 5 years prior to signing informed consent
* Patient has clinically-relevant chronic renal failure
* Patient has high blood pressure
* Patient has coronary heart disease
* Patient has known allergies to steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in OCT retinal thickness; evaluate the safety and tolerability of doses. | After 12 months of therapy.

SECONDARY OUTCOMES:
Evaluation of visual acuity; change from baseline in OCT center-point retinal thickness; the need for focal/grid laser photocoagulation during the study; the progression of diabetic retinopathy | After 12 months of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC